CLINICAL TRIAL: NCT06533995
Title: The Performance of Visuprime in Improving Ocular Surface Homeostasis and Reducing Conjunctival Bacterial Load in Patients Receiving Cataract Surgery
Brief Title: The Usefulness of Visuprime in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VF-OS-005/2021
Record Dates: First submitted 2024-07-18; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISUPRIME (Experimental): Patients receiving Visuprime eyedrop BID from Visit 1 (day -3 from surgery) to Visit 3 (day 7 from surgery).
  Interventions: Device: Visuprime
- Placebo (Placebo Comparator): Patients receiving placebo eyedrop (the vehicle of Visuprime, ie isotonic buffered saline solution) BID from Visit 1 (day -3 from surgery) to Visit 3 (day 7 from surgery).
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Visuprime — Visuprime is a medical device (class IIa sterile) with ophtalmic indication, consisting on a 10 ml multidose bottle
  Arms: VISUPRIME
Other: Placebo — placebo eyedrop isotonic buffered saline solution
  Arms: Placebo

SUMMARY:
This is a multicentre, post-market, open label, randomized, placebo-controlled prospective study exploring the performance of Visuprime in improving ocular surface homeostasis and reducing conjunctival bacterial load in patients receiving cataract surgery, as an addon treatment to postoperative standard terapy. The study will consist on 3 visits: Visit 1 (day -3 from surgery), Visit 2 (day 0, surgery), and Visit 3 (day 7 from surgery). Patients will be enrolled after having signed the informed consent form prior to any other study procedure and after inclusion/exclusion criteria check. At each visit all study procedures will be performed according to the clinical investigation plan requirements. Patients will be enrolled at Visit 1 and randomized with a 1:1 ratio to 2 groups:

GROUP A: patients receiving Visuprime eyedrop BID from day -3 to week 1. After surgery, patients will be also given standard postoperative treatment consisting on unitdose desametasone eyedrop + levofloxacin eyedrop, both given four times daily (QID) from day 0 (after surgery) to the end of the study.

GROUP B: patients receiving placebo eyedrop (the vehicle of Visuprime, i.e. isotonic buffered saline solution) BID from day -3 to week 1.

After surgery, patients will be also given standard postoperative treatment consisting on unitdose desametasone eyedrop QID + levofloxacin eyedrop QID from day 0 to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old patients, male and female
* Previous diagnosis of cataract requiring surgery
* Wishing to participate in the study and able to sign the ICF
* No topic ophthalmic medication, including lubricating eyedrops administration for at least 4 days before screening visit.

Exclusion Criteria:

* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g.rheumatic disease)
* Previous participation on this study for the fellow eye
* Increased risk of complicated cataract surgery according to the investigator assessment (for example presence of dilation less than 6 mm, pupil decentration, pseudoexfoliation, areas of iris atrophy, sublussation or lussation of the lens, complete cataract, sac instability, iridodonesis, systemic disease limiting intraoperative patient cooperation)
* Coexisting corneal diseases
* Past or active conjunctivitis - any type
* Past ocular surface burns
* Keratinization of the eyelid margin
* Sjogren syndrome
* History of corneal trauma
* Pregnant and lactating women
* Inability to self-administer study medications
* Know allergic sensitivity to any of the devices ingredients, or any other type of allergy
* Participation in a clinical trial during the 3 months prior to the beginning of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
TBUT (Tear-Break-Up-Time) | V1 (Day -3 from surgery),V2 (Day 0, surgery), V3 (Day 7 after surgery)
  To evaluate the performance of the Visuprime, used in improving ocular surface homeostasis in patients receiving cataract surgery, fluorescein tear break-up time will be measured and compared in the two groups at each visit.
TBUT (Tear-Break-Up-Time) | V3-V1 (ten days) , V2-V1(three days)
  To evaluate the performance of the Visuprime, used in improving ocular surface homeostasis in patients receiving cataract surgery, the difference in the change of Tear Break-Up Time test will be analyzed between two treatment groups at V3 compared to V1 and at V2 compared to V1.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  Ocular Surface Disease Index will be measured at each visit and compared between the two groups.
  The final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Ocular Surface Disease Index (OSDI) | V3-V1(ten days), V2-V1(three days)
  The difference in the change of Ocular Surface Disease Index will be analyzed between two treatment groups at V3 compared to V1 and V2 compared to V1.
  The final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Instantaneous Non-Invasive Break-up time (iNIBUT) | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  Instantaneous Non-Invasive Break-up time will be measured at each visit and compared between the two groups.
Instantaneous Non-Invasive Break-up time (iNIBUT) | V3-V1(ten days), V2-V1(three days)
  The difference in the change of Instantaneous Non-Invasive Break-up time will be analyzed between two treatment groups at V3 compared to V1 and V2 compared to V1.
mean Non-Invasive Break-up time (mNIBUT) | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  mean Non-Invasive Break-up time will be measured at each visit and compared between the two groups.
mNIBUT (mean NIBUT) | V3-V1(ten days), V2-V1(three days)
  The difference in the change of mean Non-Invasive Break-up time will be analyzed between two treatment groups at V3 compared to V1 and V2 compared to V1.
Tear meniscus height (TMH) | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  Tear meniscus height will be measured at each visit and compared between the two groups.
  The Tear Meniscus Height is a measurement used to assess the volume of the tear film on the ocular surface useful in diagnosing dry eye conditions.
  Tear Meniscus Height is assessed with Slit-lamp Biomicroscopy. Generally, the normal tear meniscus height is about 0.2-0.4 mm. Values below 0.2 mm often indicate a reduced tear volume, commonly associated with dry eye disease.
Tear meniscus height (TMH) | V3-V1 (ten days), V2-V1(three days)
  The difference in the change of Tear meniscus height will be analyzed between two treatment groups at V3 compared to V1 and V2 compared to V1.
  The Tear Meniscus Height is a measurement used to assess the volume of the tear film on the ocular surface useful in diagnosing dry eye conditions.
  Tear Meniscus Height is assessed with Slit-lamp Biomicroscopy. Generally, the normal tear meniscus height is about 0.2-0.4 mm. Values below 0.2 mm often indicate a reduced tear volume, commonly associated with dry eye disease.
Conjunctival hyperemia | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  Conjunctival hyperemia will be measured at each visit and compared between the two groups. This parameter will be automatically graded by Keratograph according to Efron et al.:0, normal; 1, trace; 2, mild; 3, moderate.
Corneal staining | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  Corneal staining according to Oxford Scale will be measured at each visit and compared between the two groups.
  The Oxford grading scale divides corneal staining into six groups according to severity from 0 (absent) to 5 (severe). The examiner compares the overall appearance of the patient's corneal staining with a reference figure, simulating the pattern of staining encountered in dry eye disease.
Bacterial Load | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  Conjunctival samples collected at visit 1, visit 2 and visit 3 will be analysed to determine bacterial load which will be compared in the two study groups.
VAS (Visual Analogue Scale) | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  To evaluate the safety and tolerability of the Visuprime a Visual Analogue Scale will be used for overall drop comfort and ease of instillation, with the score ranges from 0 worse to 10 better and for burning and blurred vision with the score ranges from 0 better to 10 worse. These parameters will be compared in the two groups at each visit.
5-point Likert Scale | V1 (Day -3 from surgery), V2 (Day 0, surgery), V3 (Day 7 after surgery)
  The patient satisfaction will be evaluated with a 5-point Likert Scale. The score ranges from 0 worse to 10 better.
  This parameter will be compared in the two groups at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rita Bigioni, Study Chair — not affiliated
Locations (2):
- Italy (2):
  - Policlinico Casilino, Rome, RM
  - Clinica Fabia Mater, Rome, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martucci A, Zanotto E, Curtoni A, Tiezzi Appolloni A, Corsi A. The performance of an ophthalmic solution containing Poloxamer 407 and Polyquaternium 133 in reducing conjunctival bacterial load in patients receiving cataract surgery, a randomized trial. Eur J Ophthalmol. 2025 Sep 9:11206721251375236. doi: 10.1177/11206721251375236. Online ahead of print. PMID 40924815